CLINICAL TRIAL: NCT04531813
Title: HT201307-Cumulative Irritation Patch Test (21 Day)
Brief Title: Study to Determine Skin Irritation Potential of an Antifungal Cream Containing Trolamine After Repeated Skin Application (Cumulative Irritation Patch Test)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18153
Record Dates: First submitted 2020-08-26; First posted 2020-08-31 (Actual); Results first posted 2020-09-25 (Actual); Last update posted 2020-09-25 (Actual); Status verified 2020-09

CONDITIONS: Hypersensitivity
MeSH Terms: conditions — Hypersensitivity | interventions — butenafine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Cumulative Irritation Test (Experimental): Participants received butenafine HCl 1% cream on the skin test site, 0.3% solution of sodium lauryl sulfate on the skin Positive Control test site, and a blank patch on the skin Negative Control test site daily (excluding weekends) for 21 days, or 15 applications.
  Interventions: Drug: Butenafine HCl 1% (BAY1896425); Drug: Positive Control-Sodium lauryl sulfate (SLS); Other: Negative Control

INTERVENTIONS:
Drug: Butenafine HCl 1% (BAY1896425) — Approximately 0.2 g of cream containing butenafine HCl 1% daily (excluding weekends) was applied to the absorbent pad portion of a semi-occlusive dressing, which was then applied to the skin test site. The total dose applied to each participant completing the trial was 3 g.
  Other Names: Antifungal Cream V61-044 containing Trolamine
Drug: Positive Control-Sodium lauryl sulfate (SLS) — Approximately 0.2 mL of 0.3% solution of sodium lauryl sulfate was applied to the absorbent pad portion of a semi-occlusive dressing, which was then applied to the Positive Control test site.
Other: Negative Control — A blank patch was applied to the Negative Control test site.

SUMMARY:
In this study researchers want to study the potential skin reaction after repeated application of an antifungal cream containing trolamine. The study plans to enroll about 32 healthy female or male participants with the age 18 - 79 years. Researchers will apply on the skin of the upper back between the shoulder blades of the study participants three different patches to cover a small amount of the antifungal cream or 0.3% solution of sodium lauryl sulfate, which is known to cause skin irritation (so called positive control). A third patch will cover a skin area without any product (so called negative control). Participants will return daily to the study center to have new patches containing the test products applied on the same skin area of the back, excluding weekends, for 21 days of continuous skin contact. At each visit the skin will be investigated by the researchers for redness, dryness and other reactions to learn about the skin reaction after repeated application.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have been aged 18 to 79 years, inclusive.
* Participants must have understood and executed an Informed Consent Form (ICF).
* Participants (if female) must have been willing to take a urine pregnancy test prior to the initiation and at the completion of the trial.
* Participants must have been capable of understanding and following directions.
* Participants must have been considered reliable.

Exclusion Criteria:

* Participants who were in ill health or taking medication, other than birth control, which could have influenced the purpose, integrity or outcome of the trial.
* Participants who had any visible skin disease that might have been confused with a skin reaction to the test material.
* Participants who were participating in another clinical trial at this facility or any other facility.
* Participants who were using topical or systemic steroids or antihistamines for at least 7 days prior to trial initiation and during the duration of the trial.
* Participants who had a history of adverse reaction to adhesive tape, cosmetics, over-the-counter (OTC) drugs or other personal care products.
* Participants judged by the principal investigator (PI) to be inappropriate for the trial.
* Female participants who were pregnant as evidenced by a positive urine pregnancy test, planning to become pregnant, or nursing during the course of the trial.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2013-06-10 (Actual); Primary Completion 2013-07-01 (Actual); Study Completion 2013-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Fairfield, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Undecided
Availability of this study's data will be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014. Interested researchers can use www.clinicalstudydatarequest.com to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the Study sponsors section of the portal.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was conducted at single center in the US, between 10 JUN 2013 (first subject first visit) and 1 JUL 2013 (last subject last visit).
Pre-assignment Details: A total of 32 participants were enrolled in the study and 31 received study treatment.
Period: Overall Study
Arm/Group | Cumulative Irritation Test
Started | 32
Treated | 31
Completed | 30
Not Completed | 2
Not completed — Protocol Violation | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Cumulative Irritation Test
Number analyzed (Participants) | 32
Age, Continuous [Mean (Standard Deviation); unit: Years] | 51.1 (12.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 7
Race/Ethnicity, Customized [Number; unit: Participants]
  Caucasian | 20
  Hispanic | 6
  African-American | 6

OUTCOME MEASURES:

1. Primary Outcome: Cumulative Irritation Total (CIT) Score
Description: Prior to each patch application and after the last patch removal, the test sites were evaluated for gross changes according to the Erythema Scoring Scale: 0 = No visible erythema; 0.5 = Slight, barely perceptible erythema; 1 = Mild erythema; 2 = Moderate erythema; 3 = Marked erythema; 4 = Severe erythema. The Cumulative Irritation Total is generated by totaling the Erythema Scoring Scale scores of the Investigational Product for each subject completing the trial and then adding those totals. Data is being reported for all the 30 participants as a group.
Time Frame: 21 days
Population: Subjects who received treatment and completed the study
Measure: Number; unit: Score on a scale
Arm/Group | Cumulative Irritation Test
Number analyzed (Participants) | 30
Score on a scale
  Butenafine HCl 1% | 0.0
  0.3% SLS | 20.0
  Negative Control | 0.0

ADVERSE EVENTS:
Time Frame: 21 days
Arm/Group | Cumulative Irritation Test
All-Cause Mortality (participants affected / at risk) | 0/32
Serious Adverse Events (participants affected / at risk) | 0/32
Other Adverse Events (participants affected / at risk) | 1/32
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cumulative Irritation Test (N=32)
Headache (Nervous system disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No information based on the conduct of the study (incl. protocol, data resulting from the study, or the fact that the study was being conducted) will be released without prior written consent of the sponsor unless the requirement is superseded by State or Federal law.